CLINICAL TRIAL: NCT03302780
Title: Combined Peripheral (BreEStim) and Central Electrical Stimulation (tDCS) for Neuropathic Pain Management
Brief Title: BreEStim and tDCS for Neuropathic Pain Management - Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Sheng Li, PhysicianProfessor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-14-0564 Healthy
Record Dates: First submitted 2017-10-01; First posted 2017-10-05 (Actual); Results first posted 2020-12-03 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Sham tDCS and BreEStim (Experimental): This arm includes a 20-min sham tDCS to the current dominant primary motor cortex (M1), followed by a 20-min BreEStim to the median nerve (160 times) transcutaneously on the current dominant side.
  Interventions: Device: BreEStim; Device: tDCS sham
- active tDCS (M1) and BreEStim (Experimental): This arm includes a 20-min active tDCS to the current dominant primary motor cortex (M1), followed by a 20-min BreEStim to the median nerve (160 times) transcutaneously on the current dominant side.
  Interventions: Device: BreEStim; Device: tDCS active

INTERVENTIONS:
Device: BreEStim — BreEStim will applied for 10 to 20 minutes.
Device: tDCS active — tDCS will be applied for 20 minutes.
  Arms: active tDCS (M1) and BreEStim
Device: tDCS sham
  Arms: Sham tDCS and BreEStim

SUMMARY:
This study looks at the effect of combined breathing-controlled electrical stimulation (BreEStim) and transcranial direct current stimulation (tDCS) on neuropathic pain after spinal cord injury, amputation, or brain injury. The hypothesis is that a single session of combined BreEStim and tDCS will produce an additive analgesic effect. This record covers the study in a population of healthy volunteers. Note that this study will also enroll spinal cord injury patients, brain injury patients, and amputation patients and that this study as applied to these other populations will be covered in separate ClinicalTrials.gov records.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 75 years
* male and female subjects
* healthy subjects (i.e., no recent injuries or pain)

Exclusion Criteria:

* recent injuries or pain
* have a pacemaker, or other metal and/or implanted devices
* have amputation in their arm(s)
* have spinal cord injury (SCI) involving impairment of arms
* have cognitive impairment from brain injury or are not able to follow commands, or to give consent
* have asthma or other pulmonary disease
* are not medically stable
* have preexisting psychiatric disorders
* alcohol or drug abuse
* have a history of seizures/Epilepsy, or taking benzodiazepines, anticonvulsants, and antidepressants.
* Mini-mental state examination (MMSE), a brief 30-point questionnaire test that is commonly used in the literature, will be used to screen for cognitive impairment. A brain injury patient with a score of 24 or lower on MMSE will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-04-06 (Actual); Primary Completion 2016-05-26 (Actual); Study Completion 2016-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Li, MD, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- TIRR, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham tDCS and BreEStim; Then M1 tDCS and BreEstim; M1 tDCS and BreEStim; Then Sham tDCS and BreEstim: This study has a single-blinded, single-center, sham-controlled, crossover design. It included 2 separate visits, each with either a 20-min sham tDCS or M1 tDCS to the current dominant primary motor cortex(M1), both followed by a 20-min BreEStim to the median nerve(160 times) transcutaneously on the current dominant side.
Period: Overall Study
Arm/Group | Sham tDCS and BreEStim; Then M1 tDCS and BreEstim | M1 tDCS and BreEStim; Then Sham tDCS and BreEstim
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: This study has a single-blinded, single-center, sham-controlled, crossover design. It included 2 separate visits, each with either a 20-min sham tDCS or M1 tDCS to the current dominant primary motor cortex(M1), both followed by a 20-min BreEStim to the median nerve(160 times) transcutaneously on the current dominant side.
Arm/Group | All Participants
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 34 [24 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Electrical Pain Threshold (EPT)
Description: Electrical Pain Threshold (EPT) is a type of quantitative sensory test that assesses the lowest electrical current that first evokes a sensation of pricking pain.
Time Frame: baseline, 10 minutes after tDCS, 10 minutes after BreEstim
Measure: Mean (Standard Deviation); unit: mA
Groups:
- Sham tDCS and BreEStim: This study has a single-blinded, single-center, sham-controlled, crossover design. It included a 20-min sham tDCS to the current dominant primary motor cortex(M1), followed by a 20-min BreEStim to the median nerve(160 times) transcutaneously on the current dominant side.
- Active tDCS (M1) and BreEStim: This study has a single-blinded, single-center, sham-controlled, crossover design. It included a 20-min active tDCS to the current dominant primary motor cortex(M1), followed by a 20-min BreEStim to the median nerve(160 times) transcutaneously on the current dominant side.
Arm/Group | Sham tDCS and BreEStim | Active tDCS (M1) and BreEStim
Number analyzed (Participants) | 6 | 6
mA
  Baseline | 23.83 (6.79) | 22.41 (4.67)
  After tDCS | 24.08 (7.68) | 20.41 (3.01)
  After BreEstim | 26.70 (7.68) | 23.77 (6.78)

2. Primary Outcome: Electrical Sensation Threshold (EST)
Description: Electrical Detection Threshold (EDT) is a type of Quantitative sensory test that assesses the lowest electrical current that first evokes an electrical sensation.
Time Frame: baseline, 10 minutes after tDCS, 10 minutes after BreEstim
Measure: Mean (Standard Deviation); unit: mA
Arm/Group | Sham tDCS and BreEStim | Active tDCS (M1) and BreEStim
Number analyzed (Participants) | 6 | 6
mA
  Baseline | 4.05 (1.07) | 3.54 (0.92)
  After tDCS | 3.99 (0.86) | 3.39 (0.53)
  After BreEstim | 3.95 (0.74) | 3.59 (0.64)

ADVERSE EVENTS:
Time Frame: 1 hour after treatment
Arm/Group | Sham tDCS and BreEStim | Active tDCS (M1) and BreEStim
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

LIMITATIONS AND CAVEATS:
Study stopped early, and small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No